CLINICAL TRIAL: NCT05523180
Title: A Prospective, Randomized, Double-blinded, Placebo-controlled Study Evaluating the Safety and Impact of resB® Lung Support on Quality of Life in Adult Volunteers With Chronic Obstructive Pulmonary Disease or Non-cystic Fibrosis Bronchiectasis
Brief Title: A Study to Evaluate the Effect of Probiotic Supplement on Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ResBiotic Nutrition, Inc. (Industry)
Collaborators: Nutrasource Pharmaceutical and Nutraceutical Services, Inc. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: R01-21-02-T0027
Record Dates: First submitted 2022-08-22; First posted 2022-08-31 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Chronic Obstructive Pulmonary Disease; Non-cystic Fibrosis Bronchiectasis
Keywords: COPD; NCFBE; Probiotic
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: Randomization at 1:1 ratio for active or placebo
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): 1 capsule of 15 Billion CFU proprietary probiotic blend with 120 mg herbal extracts, taken twice daily.
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): 1 capsule of placebo, taken twice daily.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — Active ingredients:
  Lactobacillus plantarum RSB11, 5 Billion colony forming units (CFU) Lactobacillus acidophilus RSB12, 5 Billion CFU Lactobacillus rhamnosus RSB13, 5 Billion CFU Holy basil leaf extract, 42.0 mg Turmeric root extract, 30.0 mg Vasaka leaf extract, 48.0 mg
  Inactive ingredients:
  Microcrystalline Cellulose, Vegan Capsule (Hypromellose), Magnesium Stearate, Silicon Dioxide
  Other Names: resB® Lung Support
  Arms: Probiotic
Other: Placebo — Active ingredients:
  N/A
  Inactive ingredients:
  Microcrystalline Cellulose, Vegan Capsule (Hypromellose), Magnesium Stearate, Silicon Dioxide
  Arms: Placebo

SUMMARY:
This study aims to evaluate the impact of a specific oral probiotic blend on the quality of life of adults with respiratory conditions.

DETAILED DESCRIPTION:
An imbalance and reduction of microbial diversity in the lung microbiota may negatively impact an individual's general health and quality of life. Further, individuals with respiratory conditions may take medications that may alter gut microbiome, which can have a negative impact on outcomes and quality of life. Evidence has emerged that there are interactions between gut and lung microbiomes, demonstrating the opportunity of using oral probiotics to support a healthy gut and/or lung microbiome, and subsequently, the general health and quality of life in this population.

ELIGIBILITY:
Inclusion Criteria:

1. Adult participants who are 18-80 years of age (inclusive).
2. Have been diagnosed with chronic obstructive pulmonary disease or non-cystic fibrosis bronchiectasis and have been on a stable treatment regimen for ≥ 6 months at screening.
3. Have a body mass index between 18.0-34.9 kg/m2 (inclusive).
4. Have normal or acceptable to the investigator vital signs (blood pressure, respiratory rate, heart rate) and normal or acceptable to the investigator physical exam findings (if applicable) at screening.
5. Individuals of childbearing potential must agree to practice a medically acceptable form of birth control for a certain time frame prior to the first dose of study product and throughout the study, including:

   1. use for at least 3 months prior to the first dose of study product: hormonal contraceptives including oral contraceptives, hormone birth control patch (e.g., Ortho Evra), vaginal contraceptive ring (e.g., NuvaRing), injectable contraceptives (e.g., Depo-Provera, Lunelle), or hormone implant (e.g., Norplant System)
   2. use for at least 1 month prior to the first dose of study product: double-barrier method, intrauterine devices, or complete abstinence from sexual intercourse that can result in pregnancy
   3. vasectomy of partner at least 6 months prior to the first dose of study product Individuals with potential to impregnate others must agree to use condom or other medically acceptable methods to prevent pregnancy throughout the study. Complete abstinence from sexual intercourse that can result in pregnancy is also acceptable.
6. Agree to refrain from treatments listed in the protocol in the defined timeframe.
7. Willing and able to agree to the requirements and restrictions of this study, be willing to give voluntary consent, be able to understand and read the questionnaires, and carry out all study-related procedures.

Exclusion Criteria:

1. Participant has a history of heart disease, uncontrolled high blood pressure (i.e., ≥160 mmHg systolic or ≥100 mmHg diastolic), renal or hepatic impairment/disease, or uncontrolled diabetes (Type I or Type II) defined as not taking a stable dose of diabetes mellitus medication on the current regimen for a minimum of three months.
2. Participants on oxygen therapy.
3. Received a vaccine for COVID-19 in the 2 weeks prior to screening or during the study period, current COVID-19 infections, or currently have the post COVID-19 condition as defined by World Health Organization (WHO) (i.e., individuals with a history of probable or confirmed SARS-CoV-2 infection, usually 3 months from the onset of COVID-19 with symptoms that last for at least 2 months and cannot be explained by an alternative diagnosis).
4. Participant has a history of unstable thyroid disease, immune disorders and/or immunocompromised (e.g. HIV/AIDS), a history of cancer (except localized skin cancer without metastases or in situ cervical cancer) within 5 years prior to screening visit.
5. Major surgery in 3 months prior to screening or planned major surgery during the course of the study.
6. Participant has consumed probiotic supplements and is unwilling to stop at least one week prior to screening and throughout the study. Supplemental probiotics may include standalone probiotic supplements, vitamins with probiotics, and any foods supplemented with probiotics.
7. Participant is currently being prescribed antibiotics or states that they have been prescribed antibiotics within the 3 months prior to screening.
8. Participant has consumed supplemental enzymes and are unwilling to stop at least one week prior to screening and throughout the study. Supplemental enzymes may include standalone enzyme supplements, probiotic supplements with enzymes, and any medications containing enzymes.
9. Participant has an abnormality or obstruction of the gastrointestinal tract precluding swallowing (e.g. dysphagia) and digestion (e.g. known intestinal malabsorption, celiac disease, inflammatory bowel disease, chronic pancreatitis).
10. Participants who are lactating, pregnant or planning to become pregnant during the study.
11. Have a known sensitivity, intolerability, or allergy to any of the study products or their excipients, or any of the rescue medications.
12. Receipt or use of an investigational product in another research study within 28 days prior to baseline visit.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2023-09-12 (Actual)

PRIMARY OUTCOMES:
To determine the effect of resB® Lung Support on quality of life | 12 weeks
  Change from baseline in St. George's Respiratory Questionnaire. The total score summarizes the impact of the condition on overall health status where 100 indicates the worst possible health status and 0 indicates best possible health status

SECONDARY OUTCOMES:
To determine the effect of resB® Lung Support on lung microbiome | 12 weeks
  Change from baseline in gut microbiome as assessed by 16S rRNA analysis from sputum samples
To determine the effect of resB® Lung Support on gut microbiome | 12 weeks
  Change from baseline in gut microbiome as assessed by 16S rRNA analysis from fecal samples
To determine the effect of resB® Lung Support on serum short-chain fatty acids | 12 weeks
  Change from baseline in serum short-chain fatty acids
To determine the effect of resB® Lung Support on stool short-chain fatty acids | 12 weeks
  Change from baseline in stool
To determine the effect of resB® Lung Support on biomarkers of inflammation | 12 weeks
  Change from baseline in serum concentration of metalloproteinase 9
To determine the effect of resB® Lung Support on biomarkers of inflammation | 12 weeks
  Change from baseline in serum concentration of tripeptide N-acetyl proline-glycine-proline
To determine the effect of resB® Lung Support on biomarkers of inflammation | 12 weeks
  Change from baseline in serum concentration of high-sensitivity C-reactive protein
To determine the effect of resB® Lung Support on biomarkers of inflammation | 12 weeks
  Change from baseline in serum concentration of pro-inflammatory cytokines
To assess the safety and tolerability of resB® Lung Support in adult participants with chronic obstructive pulmonary disease or non-cystic fibrosis bronchiectasis | 12 weeks
  Heart rate measurement
To assess the safety and tolerability of resB® Lung Support in adult participants with chronic obstructive pulmonary disease or non-cystic fibrosis bronchiectasis | 12 weeks
  Blood pressure measurement
To assess the safety and tolerability of resB® Lung Support in adult participants with chronic obstructive pulmonary disease or non-cystic fibrosis bronchiectasis | 12 weeks
  Respiratory rate measurement
To assess the safety and tolerability of resB® Lung Support in adult participants with chronic obstructive pulmonary disease or non-cystic fibrosis bronchiectasis | 12 weeks
  Weight measurement
To assess the safety and tolerability of resB® Lung Support in adult participants with chronic obstructive pulmonary disease or non-cystic fibrosis bronchiectasis | 12 weeks
  Body mass index measurement
Change in Hemoglobin levels after taking resB® Lung Support | 12 weeks
  Change in Hemoglobin levels after taking resB® Lung Support compared to baseline
Change in Mean Corpuscular Hemoglobin Concentration (MCHC) after taking resB® Lung Support | 12 weeks
  Change in Mean Corpuscular Hemoglobin Concentration (MCHC) after taking resB® Lung Support compared to baseline
Change in Albumin after taking resB® Lung Support | 12 weeks
  Change in Albumin after taking resB® Lung Support compared to baseline
Change in Total Protein after taking resB® Lung Support | 12 weeks
  Change in Total Protein after taking resB® Lung Support compared to baseline
Change in Globulin after taking resB® Lung Support | 12 weeks
  Change in Globulin after taking resB® Lung Support compared to baseline
Change in Reb Blood Cell (RBC) count after taking resB® Lung Support | 12 weeks
  Change in Reb Blood Cell (RBC) count after taking resB® Lung Support compared to baseline
Change in in Red Cell Distribution Width (RDW) after taking resB® Lung Support | 12 weeks
  Change in in Red Cell Distribution Width (RDW) after taking resB® Lung Support compared to baseline
Change in Mean Corpuscular Volume (MCV) and Mean Platelet Volume (MPV) after taking resB® Lung Support | 12 weeks
  Change in Mean Corpuscular Volume (MCV) and Mean Platelet Volume (MPV) after taking resB® Lung Support compared to baseline
Change in Mean Corpuscular Hemoglobin (MCH) after taking resB® Lung Support | 12 weeks
  Change in Mean Corpuscular Hemoglobin (MCH) after taking resB® Lung Support compared to baseline
Change in Platelet count after taking resB® Lung Support | 12 weeks
  Change in Platelet count after taking resB® Lung Support compared to baseline
Change in White Blood Cell (WBC) count after taking resB® Lung Support | 12 weeks
  Change in White Blood Cell (WBC) count after taking resB® Lung Support compared to baseline
Change in White Blood Cell (WBC) differential after taking resB® Lung Support | 12 weeks
  Change in White Blood Cell (WBC) differential after taking resB® Lung Support compared to baseline
Change in Urea after taking resB® Lung Support | 12 weeks
  Change in Urea after taking resB® Lung Support compared to baseline
Change in Sodium after taking resB® Lung Support | 12 weeks
  Change in Sodium after taking resB® Lung Support compared to baseline
Change in Potassium after taking resB® Lung Support | 12 weeks
  Change in Potassium after taking resB® Lung Support compared to baseline
Change in Chloride after taking resB® Lung Support | 12 weeks
  Change in Chloride after taking resB® Lung Support compared to baseline
Change in Creatinine after taking resB® Lung Support | 12 weeks
  Change in Creatinine after taking resB® Lung Support compared to baseline
Change in Bilirubin-total after taking resB® Lung Support | 12 weeks
  Change in Bilirubin-total after taking resB® Lung Support compared to baseline
Change in Alkaline Phosphatase after taking resB® Lung Support | 12 weeks
  Change in Alkaline Phosphatase after taking resB® Lung Support compared to baseline
Change in Aspartate Aminotransferase (AST) after taking resB® Lung Support | 12 weeks
  Change in Aspartate Aminotransferase (AST) after taking resB® Lung Support compared to baseline
Change in Alanine Aminotransferase (ALT) after taking resB® Lung Support | 12 weeks
  Change in Alanine Aminotransferase (ALT) after taking resB® Lung Support compared to baseline
Change in Estimated Glomerular Filtration Rate (eGFR) after taking resB® Lung Support | 12 weeks
  Change in Estimated Glomerular Filtration Rate (eGFR) after taking resB® Lung Support compared to baseline
Safety- participants experiencing adverse events | 12 weeks
  The number of participants experiencing Treatment Emergent Adverse Events (TEAEs)
Safety- adverse events | 12 weeks
  The total number Treatment Emergent Adverse Events (TEAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Bier, MD, Study Director — Nutrasource Pharmaceutical and Nutraceutical Services
Locations (2):
- United States (2):
  - Coral Research Clinic Corp., Miami, Florida
  - Premier Medical Associates, The Villages, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nicola T, Wenger NM, Seidman K, Evans M, Yang Y, Chen D, Van Der Pol WJ, Walia A, Lefkowitz EJ, Wang J, LeMoire A, Lin L, Morrow C, Ambalavanan N, Gaggar A, Lal CV. Double-Blind Randomized Placebo-Controlled Trial of a Lactobacillus Probiotic Blend in Chronic Obstructive Pulmonary Disease. Pulm Ther. 2025 Nov 18. doi: 10.1007/s41030-025-00333-y. Online ahead of print. PMID 41254308